CLINICAL TRIAL: NCT03374735
Title: Prospective, Multicenter, Non-controlled Study, Evaluating Safety and Performance of SETALUM™ Sealant as an add-on to Suture in Vascular Reconstruction in Patients Undergoing Carotid Enlargement Procedure Using an ePTFE Patch.
Brief Title: First In-human Use of SETALUM™ Sealant: The BlueSeal Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gecko Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GB02-CL-1401
Record Dates: First submitted 2017-12-05; First posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SETALUM™ Sealant (Experimental): SETALUM™ Sealant to be applied on the suture line
  Interventions: Device: SETALUM™ Sealant

INTERVENTIONS:
Device: SETALUM™ Sealant — SETALUM™ Sealant to be applied on the suture line

SUMMARY:
This is a prospective, multicenter, single-arm trial to evaluate the safety and performance of SETALUM™ Sealant in sealing suture lines at the anastomosis between native vessels and synthetic ePTFE vascular patch used during open vascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old;
* Surgical placement of an ePTFE patch for large carotid repair;
* Written informed consent given by the patient.

Exclusion Criteria:

* Known or suspected allergy or sensitivity to any test materials or reagents;
* Concomitant intake of immunosuppressive medications;
* Prior radiation therapy to the operating field;
* Previous surgical procedure performed on the same operating field;
* Current or recent (<3months) participation in another investigational study;
* Refusal to receive blood products;
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2017-02-07 (Actual); Study Completion 2017-10-03 (Actual)

PRIMARY OUTCOMES:
Elapsed time from clamp release to hemostasis at the suture line | During surgical procedure
  The hemostasis is observed by the operating surgeon and timed by an operative room nurse.
  Anastomotic hemostasis is defined as an anastomosis not requiring any additional intervention to control bleeding.
All adverse events occurring from the surgical procedure to Week 12 | Week 12
  Each Adverse Event was described by the seriouness and the nature of its relationship to the SETALUM™ Sealant or to the surgical procedure. The Data Monitoring Committee reviewed all occurred adverse events and provided a conclusion on the SETALUM™ Sealant safety profile.